CLINICAL TRIAL: NCT04247633
Title: Single-arm Phase II Study of Palbociclib Plus Endocrine Therapy in Patients With High Risk ER-positive/HER2-negative T1-2N0-1 Early Breast Cancer Incorporating GenesWell™ BCT
Brief Title: High Risk ER+HER2- T1-2N0-1 Early Breast Cancer With Palbociclib Plus Endocrine Therapy(HIPEx)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Collaborators: Korean Cancer Study Group (Other)
Responsible Party: Principal Investigator, Yeon Hee Park, Clinical Professor, MD, PhD, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KCSG BR19-13
Record Dates: First submitted 2020-01-27; First posted 2020-01-30 (Actual); Last update posted 2020-04-20 (Actual); Status verified 2020-04

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — palbociclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- palbociclib plus endocrine therapy treatement (Experimental): * Patients with Clinical high risk/Genomic High risk (in BCT score)-high and ER positive/HER2 negative EBC after Curative Surgery
  * Palbociclib at a dose of 125mg, orally once daily on Day 1 to Day 21 followed by 7 days off in a 28-day cycle for a total duration of 2 years
  * Standard adjuvant endocrine therapy for a duration of at least 5 years from the start of the treatment.
  Interventions: Drug: Palbociclib

INTERVENTIONS:
Drug: Palbociclib — Palbociclib at a dose of 125 mg will be administered orally once a day for 21 days, followed by 7 days off treatment of every 28 day cycle. Investigational medicinal product (IMP) will be administered with standard adjuvant endocrine therapy (Non-investigational treatment).
  Other Names: Ibrance

SUMMARY:
This is a phase II, multi-center, single-arm, open-label trial to evaluate efficacy of palbociclib with endocrine therapy as adjuvant treatment in women with C-high/G-high risk ER-positive/HER2-negative T1-2N0-1 EBC(Early Breast Cancer)

DETAILED DESCRIPTION:
The investigators hypothesized that the GenesWell™ BCT may help inform decision about whether or not to have adjuvant chemotherapy to patients with high-risk pN0-N1, ER+/HER2- breast cancer in Korea. While adjuvant therapy for ER-positive EBC is effective in reducing risk of recurrence and improving survival, recurrences are still common, especially in patients with unfavorable factors in terms of clinical, pathological and/or molecular perspectives.

Since the addition of CDK4/6 inhibitor, palbociclib, to endocrine therapy (ET) has proven clinical efficacy with tolerable toxicity profile in ER-positive, HER2-negative advanced BC, its use in the adjuvant setting may decrease risk of recurrences in patients with ER-positive, HER2-negative EBC after surgical resection of the primary tumor by enhancing primary endocrine responsiveness and preventing, or delaying the development of acquired resistance for endocrine therapy.

The purpose of this study is to evaluate the effect of addition of palbociclib to standard adjuvant ET on event-free survival (EFS) in patients with ER-positive, HER2-negative EBC but unfavorable clinicopathological (clinical high risk, C-high) and molecular features (genomic high risk, G-high).

ELIGIBILITY:
Inclusion Criteria:

1. Patient is an adult, ≥ 19 years old at the time of informed consent
2. Premenopausal and postmenopausal women or men with invasive breast cancer
3. De novo primary disease
4. Patient who performed surgery with curative aim
5. Patient who has negative surgical resection margins
6. Patient with histologically confirmed HER2-negative breast cancer
7. Patient with histologically and cytologically confirmed ER positive breast cancer by local laboratory testing
8. Pathological node assessment: pN0 or pN1
9. Tumor size ≥ 0.5 cm, and T1 or T2
10. Clinical High-Risk (Clinical high-risk patients as per the modified Adjuvant! Online guideline in the clinical trial MINADCT(Microarray in Node Negative Disease May Avoid Chemotherapy), refer to section 5.2.1)
11. Genomic High-Risk in BCT score (≥ 4)
12. Patients agreed to use effective contraception or not be of childbearing potential.
13. Patient has adequate bone marrow and organ function
14. Patient has an Eastern Cooperative Oncology Group (ECOG) performance status ≤ 1
15. Patient who is able to swallow and retain oral medication
16. A FFPE tumor sample must be available for inclusion. The tumor sample must be taken from the excised primary tumor

Exclusion Criteria:

1. Patient with recurred breast cancer
2. Patient with histologically confirmed ER negative
3. Patient with histologically confirmed HER2-positive
4. Pathological node assessment: pN2 or pN3
5. Patients has received neoadjuvant chemotherapy or endocrine therapy
6. Patient has received preoperative treatment with CDK 4/6 inhibitors.
7. Patient has received preoperative radiation therapy
8. Tumor size less than 0.5 cm
9. Patients with low clinical risk group (section 5.2.1)
10. Patients who low BCT risk group (BCT score<4)
11. Patients with lactose intolerance
12. Patients with a hypersensitivity to IP and/or components of IP
13. Pregnant women, women of childbearing potential or lactating women
14. Patients who have serious underlying co-morbidities which could cause end-organ dysfunction
15. A FFPE tumor sample is not available

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 578 (Estimated)
Dates: Start 2020-02-11 (Actual); Primary Completion 2023-02 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
3-year event-free survival | up to 3 years
  defined to be time from study entry to first event, where the first event is any type of recurrence

SECONDARY OUTCOMES:
overall survival | up to 5 years
  defined to be time from study entry to the death from any cause. Patients who lost to follow-up or have withdrawn consent to be followed will be censored at their date of last contact or withdrawal of consent to be followed, whichever occurs first.
Prognostic and predictive effects of BCT | up to 5 years
  BCT score (of GenesWell™ BCT) as a biomarker to determine the efficacy of palbociclib in combination with endocrine therapy in adjuvant setting in T1-2N0-1 high risk ER+ EBC. Performance analysis of BCT score (of GenesWell™ BCT) about predicting the effectiveness of IP.
  * BCT Score 0 - 4 (<4) :Low risk (G-low)
  * BCT score 4 - 10 (≥4) High risk (G-high)
Adverse Events | up to 2 years
  Toxicity (Adverse Events) will be collected and evaluated according to the NCI CTCAE ver. 5.0
Quality of Life (QoL) | up to 5 years
  The QoL will be evaluated using European Organization for Research and Treatment of Cancer QoL Questionnaire (EORTC QLQ-C30, and B-23)
  -These two tools for measuring quality of life were evaluated on a scale of 100 in accordance with the formula. The higher the score, the better the quality of life, and the higher the score, the more appealing the symptom scale.
Exploratory analysis of genomic biomarkers | up to 5 years
  Analysis of tumor/blood biomarker

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea